CLINICAL TRIAL: NCT06136455
Title: A Randomized Clinical Trial to Investigate Salivary Flow and pH Following Use of Essential-Oil Containing Mouthwashes
Brief Title: A Study to Investigate Salivary Flow and Potential of Hydrogen (pH) Following Use of Essential-Oil Containing Mouthwashes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCSORC005482
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Healthy
MeSH Terms: interventions — Ethanol; Mouthwashes

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Brush / Listerine Clinical Solutions Teeth Strength (Experimental): After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Clinical Solutions Teeth Strength mouthwash.
  Interventions: Drug: Listerine Clinical Solutions Teeth Strength; Drug: Colgate Cavity Protection Toothpaste
- Arm 2: Brush / Listerine Total Care Zero (Experimental): After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Total Care Zero mouthwash.
  Interventions: Drug: Listerine Total Care Zero Alcohol Mouthwash; Drug: Colgate Cavity Protection Toothpaste
- Arm 3: Brush / Listerine Cool Mint Zero (Experimental): After brushing for 1 timed minute, participants will rinse full strength for 30 seconds with Listerine Cool Mint Zero mouthwash.
  Interventions: Other: Listerine Cool Mint Zero Alcohol Mouthwash; Drug: Colgate Cavity Protection Toothpaste
- Arm 4: Brush / Water (Negative Control) (Other): After brushing for 1 timed minute, participants will rinse with for 1 minute with tap water.
  Interventions: Drug: Colgate Cavity Protection Toothpaste

INTERVENTIONS:
Drug: Listerine Clinical Solutions Teeth Strength — After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Clinical Solutions Teeth Strength mouthwash.
  Arms: Arm 1: Brush / Listerine Clinical Solutions Teeth Strength
Drug: Listerine Total Care Zero Alcohol Mouthwash — After brushing for 1 timed minute, participants will rinse full strength for 1 minute with Listerine Total Care Zero mouthwash.
  Arms: Arm 2: Brush / Listerine Total Care Zero
Other: Listerine Cool Mint Zero Alcohol Mouthwash — After brushing for 1 timed minute, participants will rinse full strength for 30 seconds with Listerine Cool Mint Zero mouthwash.
  Arms: Arm 3: Brush / Listerine Cool Mint Zero
Drug: Colgate Cavity Protection Toothpaste — Participants will brush for 1 timed minute with Colgate Cavity Protection toothpaste.

SUMMARY:
The purpose of this trial is to evaluate the amount of saliva generated and changes in the oral Potential of Hydrogen (pH) after a single use of essential oil (EO)-containing mouth rinses compared to a negative control. Three EO mouthwash formulations will be investigated in this regard, with the negative control being tap water.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and follow the requirements and restrictions of the clinical trial (including willingness to use the assigned study products per instructions, availability on scheduled visit dates and likeliness of completing the clinical trial) based upon research site personnel's assessment
* Evidence of a personally signed and dated informed consent document indicating the participant (or legally acceptable representative) has been informed of all pertinent aspects of the trial
* Able to read and understand the local language (participant is capable of reading the documents)
* Adequate oral hygiene [that is (i.e.), brush teeth daily and exhibit no signs of oral neglect]
* Adults, 18 years of age and older, in good general and oral health without any known allergy to commercial dental products or cosmetics
* Evidence of being fully vaccinated for COVID-19 (adults 60 years and older)
* Negative pregnancy urine tests (females of child-bearing potential only)
* Females of childbearing potential must be using a medically acceptable method of birth control for at least one month prior to Visit 1 and agree to continue using this method during their participation in the clinical trial
* Resting baseline unstimulated salivary sample must be equal to or greater than 0.3 mL/min to continue in the clinical trial
* A minimum of 20 natural teeth with scorable facial and lingual surfaces. Teeth that are grossly carious, extensively restored, orthodontically banded, abutments, exhibiting severe generalized cervical and/or enamel abrasion, or third molars will not be included in the tooth count
* Absence of significant oral soft tissue pathology, excluding plaque-induced gingivitis, based on a visual examination and at the discretion of the Investigator
* Absence of advanced periodontitis based on a clinical examination and discretion of the dental examiner
* Absence of fixed or removable orthodontic appliance or removable partial dentures

Exclusion Criteria:

* History of significant adverse effects, including sensitivities or suspected allergies, following use of oral hygiene products such as toothpastes, mouthwashes and red food dye
* Dental prophylaxis within four weeks prior to Visit 1
* History of medical conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures
* Use of antibiotics, anti-inflammatory or anticoagulant therapy, phenytoin sodium or diphenylhydantoin, cyclosporin A, immunostimulants/ immunomodulators during the clinical trial or within the one month prior to the Baseline exam at Visit 1. Intermittent use of certain antiinflammatory medication (ibuprofen, Aspirin); oral steroids and calcium channel blockers are acceptable at the discretion of the investigator
* Use of chemotherapeutic anti-plaque/anti-gingivitis products such as triclosan, essential oils, cetylpyridinium chloride (CPC), sodium fluoride with CPC, stannous fluoride, zinc or chlorhexidine digluconate containing mouthwashes and toothpastes within the four weeks prior to Visit 1
* Known allergy or sensitivity or history of significant adverse effects to any of the investigational product and/or product ingredients (or other ingredients in the products) specifically Cinnamyl Alcohol, Benzyl Alcohol, Citral, Citronellol, Linalool and Limonene
* Self-reported pregnancy or lactation (this criterion is due to oral tissue changes related to pregnancy and nursing which can affect interpretation of clinical trial results)
* Self-reported smokeless tobacco user including snuff, chewing tobacco, vaping and e-cigarette usage
* Males with a pregnant partner or a partner who is currently trying to become pregnant
* Suspected alcohol or substance abuse (for example, amphetamines, benzodiazepines, cocaine, marijuana, opiates)
* Significant medical or oral condition which may interfere with a participant's participation in the clinical trial, including cancer, chronic kidney disease, COPD (chronic obstructive pulmonary disease), immunocompromised state (weakened immune system) from solid organ transplant, serious heart conditions, (such as heart failure, coronary artery disease, or cardiomyopathies) Sickle cell disease, Type 2 diabetes mellitus at the discretion of the Investigator
* Participation in any clinical trial within 30 days of Visit 1
* Diagnosed Temporo-mandibular joint dysfunction/disorder
* Participants who wear bruxing devices, dental aligners, retainers
* Participants who were previously screened and ineligible or were randomized to receive investigational product
* Participants who are related to those persons involved directly or indirectly with the conduct of this clinical trial (i.e., principal investigator, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the participant inappropriate for entry into this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Salivary Flow Rate | Taken at Baseline and immediately (0), and at 2.5, 5, 10, 15, and 30 minute timepoints
  Saliva samples will be collected by participants at specified timepoints. The final amount of saliva will be weighed and flow rate will be determined.
Saliva Potential of Hydrogen (pH) | Taken at Baseline and at 2.5, 5, 10, 15, and 30 minute timepoints
  The pH value of saliva will be measured by placing the saliva sample onto the pH sensitive electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery Milleman, DDS, Principal Investigator — Salus Research, Inc.
Locations (1):
- Salus Research, Inc., Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu.